CLINICAL TRIAL: NCT06996288
Title: A Multicenter Randomized Controlled Clinical Trial of the Impact of Minimally Invasive Abdominal Surgery Esophageal Pressure Monitoring Guided Individualized PEEP on Postoperative Pulmonary Complications in Obese Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: E20241048A; E20241048A-1 (Other: TianjinCIH)
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-01

CONDITIONS: PostoperativePulmonaryComplications

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transpulmonary pressure-guided individualized PEEP group (Experimental): Preoperative assessment was performed based on basic information such as patient's age, height, weight, BMI classification, pulmonary function and blood gases. Intraoperatively, a ventilation strategy based on esophageal pressure (Pes) to monitor the transpulmonary pressure guidance was adopted, using a small tidal volume (6-8 ml/kg of ideal body weight), maintaining the transpulmonary pressure in the safe range of 5-15 cmH2O with PEEP at the level of Pes+1 cm H2O.
  Interventions: Device: Transpulmonary pressure-guided individualized PEEP
- The fixed PEEP (No Intervention): The fixed PEEP group was the intraoperative ventilation strategy based on lung protection, using a small tidal volume (6-8 ml/kg of ideal body weight) and setting the PEEP level at 8 cmH2O.

INTERVENTIONS:
Device: Transpulmonary pressure-guided individualized PEEP — Transpulmonary pressure-guided individualized PEEP group was an intraoperative ventilation strategy based on esophageal pressure (Pes) monitoring of transpulmonary pressure-guided ventilation, using a small tidal volume (6-8 ml/kg of ideal body weight), maintaining the transpulmonary pressure in the safe range of 5-15 cmH2O PEEP for Pes+1 cm H2O level.
  Arms: Transpulmonary pressure-guided individualized PEEP group

SUMMARY:
The aim of this study is to compare the effect of individualized PEEP based on transmural lung pressure and fixed PEEP on postoperative pulmonary complications during laparoscopic or robotic abdominal surgery in obese patients.

The main questions are:

1. whether the intraoperative application of individualized PEEP in obese patients can reduce the incidence of postoperative pulmonary complications at 7d, 30d, and 90d postoperatively compared to fixed PEEP
2. Whether the application of individualized PEEP in obese patients can optimize intraoperative respiratory mechanics, oxygenation index (PaO2/FiO2), PaCO2, and EtCO2 compared with fixed PEEP.

3 Whether the application of individualized PEEP in obese patients can reduce the incidence of non-respiratory complications, postoperative QoR-15 scores, unplanned reintubation, unplanned transfers, and unplanned extubation in the postoperative period compared with fixed PEEP. planned reintubation, unplanned transfers to ICU and ICU days, hospitalization days, 30-day and 90-day mortality.

Participants will:

Patients with BMI >= 30 kg/m² undergoing laparoscopic or robotic abdominal surgery received PEEP during surgery (divided into individualized PEEP and fixed PEEP), and were followed up for 90 days to observe the incidence of pulmonary complications and related study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age; ASA class I-III. Patients undergoing bariatric laparoscopic or robotic abdominal surgery; BMI ≥30 kg/m²; Planned operative time ≥120 minutes.

Exclusion Criteria:

- Presence of other serious cardiorespiratory diseases, such as severe chronic obstructive pulmonary disease (COPD, GOLD Class III-IV); history of severe or uncontrolled bronchial asthma, history of pulmonary resection; Presence of unstable cardiovascular disease, NYHA classification 3-4, such as severe arrhythmias or heart failure; Presence of neuromuscular disease affecting respiratory function, such as severe spinal cord injury; intracranial injury history of esophageal-related surgery, contraindications to esophageal catheter insertion, including severe coagulopathy (platelets < 5000/μL or INR > 4) severe chronic liver disease (Child-Pugh score ≥ 12) Patients who cannot be extubated in time after surgery and need to return to the ICU with an endotracheal tube or are scheduled to be reintubated after surgery.

(7) general anesthesia duration less than 120 minutes

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
PostoperativePulmonaryComplications | From enrollment to seven days postoperatively
  The primary outcome was acomposite of pulmonary complications within the first 7 postoperative days, including respiratory failure, acute respiratory distress syndrome, bronchospasm, new pulmonaryinfiltrates, pulmonary infection, aspiration pneumonitis, pleural effusion, atelectasis, cardiopulmonary edema, and pneumothorax.